CLINICAL TRIAL: NCT05525832
Title: Effect of Nasopharyngeal Wash With Normal Saline on SARS-CoV2 Viral Load: A Randomized Controlled Trial
Brief Title: Effect of Nasopharyngeal Wash With Normal Saline on SARS-CoV2 Viral Load
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Larissa University Hospital (Other)
Responsible Party: Principal Investigator, Ioannis Pantazopoulos, Assistant Professor of Emergency Medicine, Larissa University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 13148
Record Dates: First submitted 2022-08-26; First posted 2022-09-02 (Actual); Last update posted 2022-09-02 (Actual); Status verified 2022-08

CONDITIONS: SARS-CoV2 Infection
Keywords: Nasopharyngeal wash; Normal saline; SARS-CoV2; Viral load
MeSH Terms: conditions — COVID-19 | interventions — Saline Solution; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Randomized Pilot Controlled Trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Normal saline group (Experimental): Patients that will receive normal saline 0.9% solution for nasopharyngeal wash
  Interventions: Other: Normal saline
- control group (No Intervention): Patients that will not perform nasopharyngeal washes

INTERVENTIONS:
Other: Normal saline — Nasopharyngeal washes with NaCl 0.9%
  Other Names: NaCl 0.9%
  Arms: Normal saline group

SUMMARY:
Although great progress has been made over the past 2 years in the scientific understanding of the biology, epidemiology, and pathogenesis of severe acute respiratory syndrome coronavirus 2 (SARS-CoV2), case morbidity and fatality rates remain a great concern and continue to challenge the healthcare resources worldwide as novel variants emerge. There is therefore an urgent need for affordable and readily available strategies to reduce viral transmission. Previous studies in non coronavirus disease 2019 (COVID-19) patients have demonstrated that administration of low-salt (isotonic but 0.0375% Na) and isotonic saline (0.9% Na) solutions has been associated with an immediate, significant reduction in the microbial antigens and a related decline of microbial burden. The primary aim of the present study is to determine the effect of nasal washes with normal saline 0.9% on nasopharyngeal viral load in hospitalized patients with COVID-19 pneumonia. The secondary aim is to examine if this effect influences escalation to high flow nasal oxygen or non-invasive ventilation and admission to ICU in patients with COVID-19 pneumonia.

DETAILED DESCRIPTION:
Investigators will perform a prospective, randomized, pilot, controlled study in 50 patients with confirmed COVID-19 pneumonia. All patients will be treated with the standard protocol of care for COVID-19 at the Department of Infectious Diseases and will be randomized into one of two groups with the method of sequentially numbered, opaque, sealed envelopes, the normal saline group (will receive normal saline 0.9% solution for nasopharyngeal wash) and the control group (no treatment). In all patients, an initial baseline nasopharyngeal swab will be obtained at admission and will be placed in a sterile bottle of virus transport medium for SARS-CoV2 nucleic acid detection (day 1). Then, an educational review of nasopharyngeal wash technique will be performed. Patients from the normal saline group will be provided with eight 10 mL sterile bottles of sodium chloride 0.9% (NaCl 0.9%) solution and will be advised to perform nasopharyngeal wash with 10 ml of solution to each nostril, every 4 hours for a 16-hour period. Twenty-four hours after the baseline nasopharyngeal swab, and 8 hours after the last nasopharyngeal wash, a second nasopharyngeal swab will be collected for measurement of the viral load (day 2). All nasopharyngeal swabs will be collected by a physician blinded to group allocation and will be collected from the same nostril for each patient. Each sample will be tested at most up to 12 hours following collection. Patients demographic and clinical information will be recorded at admission [need for escalation to high flow nasal cannula (HFNC) or non invasive ventilation (NIV). Disease-related symptoms and potential adverse effects related to use of normal saline will also be monitored. All patients will be followed until hospital discharge, intensive care unit (ICU) admission or death. Those that will be discharged will be reexamined 14 days after hospital discharge for real-time polymerase chain reaction (RT-PCR). Manual chart review will be used to gather details of the laboratory studies, course, and outcomes.

ELIGIBILITY:
Inclusion Criteria:

* adult patients hospitalized primarily for COVID-19 pneumonia
* confirmed SARS-CoV2 infection diagnosed through RT-PCR test of nasopharyngeal samples

Exclusion Criteria:

* patients with confirmed SARS-CoV2 infection who were not primarily admitted for COVID-19 pneumonia
* patients with use of intranasal sprays for at least two weeks prior to study enrollment
* sinonasal surgery within 3 months prior to study enrollment
* patients with sinusitis
* inability to perform nasopharyngeal wash
* participation in other trials

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
SARS-CoV2 viral load | 24 hours
  SARS-CoV2 viral load in nasopharyngeal swab in hospitalized patients with COVID-19 pneumonia

SECONDARY OUTCOMES:
Need for escalation to HFNC / NIV, ICU admission | From date of randomization until hospital discharge, ICU admission or date of death from any cause, whichever came first assessed up to 3 months
  Number of participants with need for escalation to high flow nasal oxygen or non-invasive ventilation or ICU admission in patients with COVID-19 pneumonia.

CONTACTS AND LOCATIONS:
Overall Officials: Ioannis Pantazopoulos, MD, Study Director — University Hospital of Larissa
Locations (1):
- University Hospital of Larissa, Larissa, Thessaly, Greece

IPD SHARING:
Plan to Share IPD: Yes
all collected individual participant data (IPD)
Time Frame: For one year after the end of the study
Access Criteria: Contact study director by e-mail

REFERENCES:
- [Background] Petersen E, Ntoumi F, Hui DS, Abubakar A, Kramer LD, Obiero C, Tambyah PA, Blumberg L, Yapi R, Al-Abri S, Pinto TCA, Yeboah-Manu D, Haider N, Asogun D, Velavan TP, Kapata N, Bates M, Ansumana R, Montaldo C, Mucheleng'anga L, Tembo J, Mwaba P, Himwaze CM, Hamid MMA, Mfinanga S, Mboera L, Raj T, Aklillu E, Veas F, Edwards S, Kaleebu P, McHugh TD, Chakaya J, Nyirenda T, Bockarie M, Nyasulu PS, Wejse C, Muyembe-Tamfum JJ, Azhar EI, Maeurer M, Nachega JB, Kock R, Ippolito G, Zumla A. Emergence of new SARS-CoV-2 Variant of Concern Omicron (B.1.1.529) - highlights Africa's research capabilities, but exposes major knowledge gaps, inequities of vaccine distribution, inadequacies in global COVID-19 response and control efforts. Int J Infect Dis. 2022 Jan;114:268-272. doi: 10.1016/j.ijid.2021.11.040. Epub 2021 Dec 1. No abstract available. PMID 34863925
- [Background] Zou L, Ruan F, Huang M, Liang L, Huang H, Hong Z, Yu J, Kang M, Song Y, Xia J, Guo Q, Song T, He J, Yen HL, Peiris M, Wu J. SARS-CoV-2 Viral Load in Upper Respiratory Specimens of Infected Patients. N Engl J Med. 2020 Mar 19;382(12):1177-1179. doi: 10.1056/NEJMc2001737. Epub 2020 Feb 19. No abstract available. PMID 32074444
- [Background] Jajou R, Mutsaers-van Oudheusden A, Verweij JJ, Rietveld A, Murk JL. SARS-CoV-2 transmitters have more than three times higher viral loads than non-transmitters - Practical use of viral load for disease control. J Clin Virol. 2022 Jun;150-151:105131. doi: 10.1016/j.jcv.2022.105131. Epub 2022 Mar 14. PMID 35395500
- [Background] Pujadas E, Chaudhry F, McBride R, Richter F, Zhao S, Wajnberg A, Nadkarni G, Glicksberg BS, Houldsworth J, Cordon-Cardo C. SARS-CoV-2 viral load predicts COVID-19 mortality. Lancet Respir Med. 2020 Sep;8(9):e70. doi: 10.1016/S2213-2600(20)30354-4. Epub 2020 Aug 6. No abstract available. PMID 32771081
- [Background] Rabaan AA, Tirupathi R, Sule AA, Aldali J, Mutair AA, Alhumaid S, Muzaheed, Gupta N, Koritala T, Adhikari R, Bilal M, Dhawan M, Tiwari R, Mitra S, Emran TB, Dhama K. Viral Dynamics and Real-Time RT-PCR Ct Values Correlation with Disease Severity in COVID-19. Diagnostics (Basel). 2021 Jun 15;11(6):1091. doi: 10.3390/diagnostics11061091. PMID 34203738
- [Background] Tom MR, Mina MJ. To Interpret the SARS-CoV-2 Test, Consider the Cycle Threshold Value. Clin Infect Dis. 2020 Nov 19;71(16):2252-2254. doi: 10.1093/cid/ciaa619. No abstract available. PMID 32435816
- [Background] Huijghebaert S, Hoste L, Vanham G. Correction to: Essentials in saline pharmacology for nasal or respiratory hygiene in times of COVID-19. Eur J Clin Pharmacol. 2021 Sep;77(9):1295. doi: 10.1007/s00228-021-03141-w. No abstract available. PMID 33893861